CLINICAL TRIAL: NCT00123396
Title: VHA Clinicians and Bioterror Events: Interactive Web-based Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BTI 02-092
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Smallpox; Anthrax
Keywords: Bioterrorism; Education, Medical, Continuing; Internet
MeSH Terms: conditions — Smallpox; Anthrax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Test the effectiveness of the BioCASES teaching modules by way of a randomized controlled trial of VAMCs using the BioTESTS to evaluate their effectiveness for increasing and sustaining VA clinician knowledge, skills, and ability to respond to bioterrorism events.
  Interventions: Behavioral: BioCASES and BioTESTS

INTERVENTIONS:
Behavioral: BioCASES and BioTESTS

SUMMARY:
Our 4-year project uses public domain software and content developed by a University of Alabama at Birmingham (UAB) team and updates, refines, and tailors it to the unique clinician populations and electronic educational applications of VAMCs We are testing an innovative, web-based intervention adapted specifically for the VA to increase syndromic recognition, treatment, and post-exposure prophylaxis of biological warfare agents at multiple VA sites via a randomized controlled trial (RCT). Ultimately, we will disseminate the intervention throughout the entire VA system.

DETAILED DESCRIPTION:
Background:

Because of VA's long history in disaster preparedness, and the crucial role VA providers will play, the VA medical system has the potential to make an enormous difference in outcomes following a bioterror attack or infectious outbreak. A 2002 AHRQ report reviewed 60 studies and found that very few bioterrorism preparedness training programs were rigorously evaluated. Our project was the first effort to formally test and implement a bioterrorism preparedness intervention in the VA healthcare system. Because Internet-delivered interventions have the potential for wide dissemination, we used the Internet to implement the Intervention.

Objectives:

1. To develop, tailor, and continuously update and validate evidence- and scenario-based electronic teaching and testing modules to increase VA clinicians' knowledge of Category A biological warfare agents. We refer to these instruments as Bioterrorism Case Analysis and Skills Enhancement Sessions (BioCASES) and Bioterrorism Skills Test Sessions (BioTESTS).
2. To test the effectiveness of the BioCASES teaching modules by way of a randomized controlled trial of VAMCs using the BioTESTS to evaluate their effectiveness for increasing and sustaining VA clinician knowledge, skills, and ability to respond to bioterrorism events.
3. To continue to develop and adapt BioCASES and BioTESTS for use in VA CME programs. Ultimately, we will disseminate the intervention throughout the entire VA system.

Methods:

Our project team developed or refined and updated a total of 12 educational modules focusing on CDC's Category A agents and other emerging infectious diseases. We developed post-test instruments and case-based scenarios germane to the VA patient population for anthrax and smallpox. Materials were designed specifically for the unique clinician populations and electronic educational applications available in VAMCs. Website functionality and content were refined using the nominal group technique and "thinking aloud" protocols. We tested our innovative, web-based educational intervention at fifteen VA facilities via a randomized controlled trial (RCT).

Status:

The intervention has been completed. Fifteen sites were randomized and completed the study processes.

ELIGIBILITY:
Inclusion Criteria:

Clinicians at participating facilities who work in a primary care setting (ED, MOD, general medicine, primary care, or CBOC).

Exclusion Criteria:

Facilities will be excluded from the project that 1)choose not to participate, or 2)do not have the minimum number of clinicians needed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-08; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The outcome measure will be performance on post-test administered immediately and at 3 months and 6 months post intervention. Performance on the post-test administered at three months will be considered the main outcome of the study. | 3 months

SECONDARY OUTCOMES:
The 6-month tests will be given to demonstrate the sustainability of the intervention (prevention of decay effect).

CONTACTS AND LOCATIONS:
Overall Officials: Catarina I. Kiefe, PhD MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL; Thomas K Houston, MD MPH, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (9):
- United States (9):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

REFERENCES:
- [Result] Abdolrasulnia M, Strasser S, Pryor E, Terndrup T, Weissman NW, Williams M, Heck E, Casebeer L. Spatial Patterns Representing the Geographic Impact of Physician Participation in an Online CME Bioterrorism Course Following the Anthrax Events of 2001. Medinfo. 2004 Dec 1; 2004(CD):1498.
- [Result] Bennett NL, Casebeer LL, Kristofco RE, Strasser SM. Physicians' Internet information-seeking behaviors. J Contin Educ Health Prof. 2004 Winter;24(1):31-8. doi: 10.1002/chp.1340240106. PMID 15069910
- [Result] Terndrup T, Nafziger S, Weissman N, Casebeer L, Pryor E. Online bioterrorism continuing medical education: development and preliminary testing. Acad Emerg Med. 2005 Jan;12(1):45-50. doi: 10.1197/j.aem.2004.08.040. PMID 15635137
- [Result] O'Byrne WT, Terndrup TE, Kiefe CI, Weissman NW. A Primer on Biological Weapons for the Clinician, Part I. Johns Hopkins Advanced Studies in Medicine. 2003 Feb 1; 3:75-86.
- [Result] O'Byrne WT, Terndrup TE, Kiefe CI, Weissman NW. A Primer on Biological Weapons for the Clinician, Part II. Johns Hopkins Advanced Studies in Medicine. 2003 Mar 1; 3:157-167.
- [Result] Casebeer LL, Strasser SM, Spettell CM, Wall TC, Weissman N, Ray MN, Allison JJ. Designing tailored Web-based instruction to improve practicing physicians' preventive practices. J Med Internet Res. 2003 Jul-Sep;5(3):e20. doi: 10.2196/jmir.5.3.e20. Epub 2003 Sep 25. PMID 14517111
- [Result] Filoromo C, Macrina D, Pryor E, Terndrup T, McNutt SD. An innovative approach to training hospital-based clinicians for bioterrorist attacks. Am J Infect Control. 2003 Dec;31(8):511-4. doi: 10.1016/s0196-6553(03)00699-0. PMID 14647116